CLINICAL TRIAL: NCT05026671
Title: The Effect of The Use of a Videolaryngoscope and/or Stylet on Intubation Time in Obese Patients: A Randomized Clinical Trial
Brief Title: The Effect of The Use of a Videolaryngoscope and/or Stylet on Intubation Time in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-2021/04
Record Dates: First submitted 2021-08-22; First posted 2021-08-30 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2021-08

CONDITIONS: Intubation Time
Keywords: Obese Patients; Stylet Procedures; Video Laryngoscope; First-attempt intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and the healthcare worker who will perform preoperative and postoperative visit will be blinded to randomized study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group DL (Active Comparator): The control group consists of intubating the trachea with an endotracheal tube alone (without stylet).
  Interventions: Procedure: Endotracheal Tube Alone
- Group DLS (Experimental): The Experimental group consists of intubating the trachea with an endotracheal tube + stylet.
  Interventions: Procedure: Endotracheal Tube+ Stylet
- Group VL (Experimental): The Experimental consists of intubating the trachea with an endotracheal tube + Video-laryngoscope
  Interventions: Procedure: Endotracheal Tube + Video-laryngoscope
- Group VLS (Experimental): The Experimental consists of intubating the trachea with an endotracheal tube + stylet + Video-laryngoscope
  Interventions: Procedure: Endotracheal tube + stylet with Video-laryngoscope

INTERVENTIONS:
Procedure: Endotracheal Tube Alone — Intubating the trachea with an endotracheal tube alone ( without stylet).
  Arms: Group DL
Procedure: Endotracheal Tube+ Stylet — Intubating the trachea with an endotracheal tube + stylet.
  Arms: Group DLS
Procedure: Endotracheal Tube + Video-laryngoscope — Intubating the trachea with an endotracheal tube + Video- laryngoscope
  Arms: Group VL
Procedure: Endotracheal tube + stylet with Video-laryngoscope — Intubating the trachea with an endotracheal tube + stylet + Video-laryngoscope
  Arms: Group VLS

SUMMARY:
Although many researchers would agree that obesity per se is not a risk factor for difficult intubation, there are many well known obesity-related challenges in airway management including difficulty with mask ventilation, more frequent and rapid oxygen desaturation, increased oxygen consumption, and increased sensitivity to the respiratory depressant effects of anesthetic and analgesic drugs. Hence, in these conditions, rapid and nontraumatic intubation gain higher interest. There is controversy about using videoaryngoscopy (VL) in obese patients in these difficult situations. The primary aim of this study is to compare, in terms of intubation time, VL,VL plus stylet and direct-laryngoscopy(DL) plus stylet combination with DL alone in obese patients.

DETAILED DESCRIPTION:
Patients who will be scheduled for surgeries requiring endotracheal intubation, with a body mass index (BMI) more than 30 kg/m2, will be included to this study. During preanesthetic visit (performed by an anesthesiologist not involved in this study) history of difficult intubation, measurement of common predictive indices for difficult intubation (BMI, thyromental distance, neck circumference, Mallampati grade, interincisal [or intergingival] distances), and evaluation of status of dentition and neck movement will be noted.

In the operating room, all patients will be connected to standard monitoring devices. Anesthesia induction will be carried out according to our hospital obese patient anesthesia management protocol. Then, after induction of anesthesia, the patients will be intubated one of four pre-defined protocols that will be determined via randomization during a preanesthetic visit by a person who is unfamiliar with the research protocol.

Primary hypothesis of this study is; using a video-laryngoscope plus stylet will reduce the time required to achieve successful tracheal intubation in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented body mass index (BMI) of ≥ 30.
* Patients scheduled to undergo inpatient surgery procedures under general anesthesia.
* Willingness and ability to sign an informed consent document 18 - 80 years of age

Exclusion Criteria:

* Patients who are deemed to be such a significant of an airway risk that they necessitate awake fiberoptic intubation
* Patients with a history of facial abnormalities, oral-pharyngeal cancer, or reconstructive surgery
* Emergency surgeries
* Pregnancy
* Any other conditions or use of any medication which may interfere with the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Intubation Time Using a Stop Watch | Up to 3 minutes
  The timing measurements will begin once the laryngoscope blade will be placed in the patient's mouth and ended when an end-tidal CO2 tracing will be detected.

SECONDARY OUTCOMES:
Heart Rate | Before induction to 3 min after intubation
  Before induction, after induction, after intubation, after intubation at 1st minute, 2nd minute, and 3rd minute
Mean Arterial Pressure: | Before induction to 3 min after intubation
  Before induction, after induction, after intubation, after intubation at 1st minute, 2nd minute, and 3rd minute
Saturation | Before induction to 3 min after intubation
  Before induction, after induction, after intubation, after intubation at 1st minute, 2nd minute, and 3rd minute
Incidence of severe complications following intubation | During intubation to 3 min after intubation
  Hypoxia, collapse, cardiac arrest, death.
Glottis View Using the Cormack Lehane Score | Up to 1 minute
  Cormack Lehane score classification
  Grade 1: Most of the glottis is visible Grade 2: At best almost half of the glottis is seen, at worst only the posterior tip of the arytenoids is seen Grade 3: Only the epiglottis is visible Grade 4: No laryngeal structures are visible
Glottis View Using the POGO Score | Up to 1 minute
  the POGO score evaluate the glottic view during tracheal intubation using a classification of 1/2/3/4 and a score of 0% to 100%, respectively. The POGO score denote visualization of the entire glottic opening from the anterior commissure to the posterior cartilages, and a score of 0% denotes inability to visualize any part of the glottic opening.
Number of intubation attempts | Up to postinduction 120 second
  An intubation attempt will be defined as the insertion of the laryngoscope blade into the mouth of the patient, regardless of whether an attempt will be made to insert a tracheal tube. More than 5 attempts or 120 s will be regarded as a failure of intubation.
Ease of Intubation | Up to 1 minute
  Subjective evaluation of the anesthesiologist, rated as (1) very easy, (2) easy, (3) moderate, (4) difficult, and (5) impossible.
Complications related to intubation | postoperative 4th hour
  A postoperative follow-up assessment will be performed approximately 4 hr after surgery by a co-investigator blinded to the intubation device to evaluate the presence and severity of sore throat, any changes in voice, trauma to the lip, tongue, gum, or teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD, DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)